CLINICAL TRIAL: NCT06797258
Title: Safety And Effectiveness Of FlexHD® Pliable Acellular Dermal Matrix In Implant-Based Breast Reconstruction
Brief Title: FlexHD® Pliable Investigation in Implant-Based Breast Reconstruction
Acronym: SHAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Collaborators: MCRA (an IQVIA business) (Unknown); Bruder Consulting International, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTF 2024-10-IDE
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Implant Based Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): FlexHD® Pliable
  Interventions: Device: FlexHD® Pliable; Other: No intervention

INTERVENTIONS:
Device: FlexHD® Pliable — Acellular Dermal Matrix
Other: No intervention — Historical Control Arm

SUMMARY:
Prospective, multi-center, single-arm clinical study in females undergoing immediate implant-based breast reconstruction using a pre-pectoral technique

ELIGIBILITY:
Inclusion Criteria:

* Females at least 22 years of age
* Scheduled to undergo unilateral or bilateral mastectomy with immediate implant-based, prepectoral breast reconstruction
* Willing to provide Informed Consent
* Able to return for all required study visits
* Must read and understand English language

Exclusion Criteria:

* Is of childbearing potential and has a positive pregnancy test within 7 days of study procedure
* Has a residual gross tumor at the intended reconstruction site
* Has undergone previous breast surgery, such as lumpectomy or breast augmentation, at the site of implantation with the exception of a biopsy
* Has undergone previous radiation therapy to the reconstruction site or chest wall, or is scheduled to undergo post-operative radiation therapy at the reconstruction site
* Completed chemotherapy within 3 weeks prior to surgery
* Has been diagnosed with a comorbid condition determined by the investigator to place the subject at an increased risk of complications
* Has a Body Mass Index (BMI) >35
* Has used nicotine products within 1 month of screening
* Must not have taken oral corticosteroids for a minimum of 1 month prior to the procedure or have a history of long-term use of systemic oral corticosteroids or anticipate the use during course of the study

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of major complication | 12 months
  Complications that require additional hospitalization or reoperation
Frequency of reconstructive failure | 12 months
  Removal/explantation of the breast implant

SECONDARY OUTCOMES:
Change in patient reported outcomes | 12 months
  Change from baseline in patient reported outcomes as measured by the BREAST-Q (Scoring 0-100; 0=less satisfaction; 100= greater satisfaction)
Pain | 12 months
  Pain scores as measured by the Numerical Pain Rating Scale (NPRS) (Scoring 0-10; 0=no pain; 10= worst imaginable pain)
Adverse events | 12 months
  Reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Jonathan Heistein, MD Plastic & Reconstructive Surgery, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No